CLINICAL TRIAL: NCT05529433
Title: Pain Assessment During Chemo-Mechanical and Smart Burs Caries Removal Versus Atraumatic Restorative Treatment in Carious Primary Molars: A Randomized Clinical Trial
Brief Title: Pain Assessment During Chemo-Mechanical and Smart Burs Caries Removal Versus Atraumatic Restorative Treatment in Carious Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Mahmoud Abdel Sattar El sayed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: b9xe7bsh
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atraumatic Restorative Treatment (ART) (Active Comparator): Atraumatic Restorative Treatment is a simple technique based on preservation of sound tooth structure and minimal patient's discomfort.
  Interventions: Procedure: Atraumatic Restorative Treatment (ART)
- Smart Burs (Experimental): Smart Burs are minimally invasive technique which selectively removes the infected carious dentin leaving the affected intact dentin.
  Interventions: Procedure: Smart Burs
- Chemo-Mechanical Caries Removal (CMCR) (Experimental): A chemical agent which selectively removes the carious dentin by breaking the denatured collagen fibers making them soft and preserving the healthy dentin without drilling.
  Interventions: Procedure: Chemo-Mechanical Caries Removal (CMCR)

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment (ART) — Atraumatic Restorative Treatment is highly accepted by the patients as there is no need for local anesthesia. It is a minimal invasive technique which preserves sound tooth structure as caries removal will be done by a sharp spoon excavator. It requires less time during caries removal. There is a chemical bond between the tooth and the glass ionomer adhesive material. So, there is no need for cutting sound tooth structure for retention of the restoration.
  Arms: Atraumatic Restorative Treatment (ART)
Procedure: Smart Burs — Smart Bur is a polymer bur which removes only soft infected dentin as the cutting edges become dull in contact with the hard affected dentin.Caries removal will be done by Smart Bur mounted on a low speed hand-piece leaving the affected dentin intact. It requires less time for caries removal.
  Arms: Smart Burs
Procedure: Chemo-Mechanical Caries Removal (CMCR) — Selecti-Solve gel is a dental gel which main active ingredient is Papain enzyme which selectively removes the caries without pain and has bacteriostatic, bactericidal and anti-inflammatory properties. The use of CMCR is recommended as an alternative treatment technique in anxious patients. The gel will be applied with a blunt spoon instrument and distributed well into the cavity according to manufacturer's instructions.
  Other Names: Selecti-Solve gel (Denta Pharma, Egypt)
  Arms: Chemo-Mechanical Caries Removal (CMCR)

SUMMARY:
The aim of the clinical trial is to assess pain during Atraumatic Restorative Treatment (ART), Smart Burs and Chemo-mechanical Caries Removal (CMCR) in primary molars.

DETAILED DESCRIPTION:
The principles of the caries removal have changed greatly in the last decade. The use of local anesthesia with conventional techniques"high-speed hand piece" increase the fear and anxiety of the child. Minimally invasive techniques reduce the pain and anxiety of the child by eliminating the use of local anesthesia.

In ART, soft carious tissue is removed by hand instruments. Although this technique is very simple.

Moreover, Smart Burs are more efficient in removal of soft infected dentine than ART leaving the affected dentin intact; as when they touch hard dentin, they become dull.

Finally, the recent effective method of caries removal is CMCR. The chemical agent contains proteolytic enzyme which destructs partially degraded collagen, leaving the infected dentin soft and easy to be excavated.

Therefore, the aim of this study is to assess pain during Atraumatic Restorative treatment, Smart Burs and Chemo-Mechanical Caries Removal in primary molars.

ELIGIBILITY:
Inclusion Criteria:

* Caries in second primary molars within enamel/ dentin without pulp disease.
* There is a clear band of dentin coronal.
* Cooperative and healthy children.

Exclusion Criteria:

* Presence of signs and symptoms of necrosis.
* Root caries.
* History of spontaneous pain.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | at baseline
  The pain will be assessed by Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Time taken for caries removal | at baseline
  The time is measured by a stopwatch in minutes
Efficacy of caries removal | at baseline
  The efficacy of caries removal will be assessed by Caries Detector dye.

CONTACTS AND LOCATIONS:
Overall Officials: Rania Nasr, Professor, Study Director — Cairo University; Rasha Hatem, Associate Professor, Study Director — Cairo University; Reham Mahmoud, BDS, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided